CLINICAL TRIAL: NCT06746974
Title: Comparing the Effects of Extracorporeal Shockwave Therapy and Splinting in the Treatment of Trigger Finger
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2024/819
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Trigger Finger; Shockwave Therapy
Keywords: trigger finger; shockwave
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Splints

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave (Experimental)
  Interventions: Device: Shockwave
- Splint (Active Comparator)
  Interventions: Device: Splint

INTERVENTIONS:
Device: Shockwave — In the Shockwave group, will be applied focused shockwaves therapy of 1500 impulses at 0.01 mJ/mm2 over the painful area or the pathologic flexor tendon to each participant under the supervision of a physiatrist. The ESWT will be conducted once weekly for 4 weeks with a sham splint (DIP joint blocking splints) for at least 8 hours per day for 6 weeks.
  Arms: Shockwave
Device: Splint — In the splinting group, will be provided a PIP blocking splint at least 8 hours per day for 6 weeks with the sham shockwave (the patients close their eyes, extend their hand through a partition, apply shockwave device head with gel on the patient's finger, and play a mobile phone sound that mimics the sound of a real shockwave machine) once a week for 4 weeks.
  Arms: Splint

SUMMARY:
The goal of this study is to compare the effects of extracorporeal shockwave therapy and splinting in the treatment of trigger finger.

Participants will:

Be randomized into two groups (shockwave group and splint group). Visit the clinic once a week for four weeks for therapy. Keep a diary of their symptoms, which will be reviewed at six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years
* Grade I-III trigger finger patients (patients who has the presence of tenderness over the A1 pulley or painful locking or triggering as they fixed and extended the finger)
* Patients who consented to participation in the study

Exclusion Criteria:

* Trigger thumb
* The patients who had received previous treatment (steroid injection, ESWT or surgical release)
* Patients with local infections, malignancies, severe coagulopathy and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
100-mm. horizontal VAS score | at enrollment, fourth week, and sixth week after first intervention
  The VAS or Visual Analog Scale is a scale that is used to evaluate the level of pain. It is represented by a horizontal line that is 100-mm. long. The score is determined by measuring the distance in mm. A higher score on this scale indicates greater pain intensity.

SECONDARY OUTCOMES:
QuickDASH score | at enrollment, fourth week, and sixth week after first intervention
  The QuickDASH or Quick Disabilities of the Arm, Shoulder and Hand is a questionnaire that is used to evaluate the ability to perform activities of the arm, shoulder, and hand. It consists of 11 questions that patients are required to answer all of them. The answers are summarized in a range of 0-100, where a higher score indicates greater disability.
Number of triggering | at enrollment, fourth week, and sixth week after first intervention
  The number of triggering events in ten active full fists will be scored out of ten. If a participant's finger remain locked at any time in making ten active full fists, they will be asked to stop and given a score of 10/10

IPD SHARING:
Plan to Share IPD: No
Due to concerns about patient privacy, confidentiality, and ethical obligations

REFERENCES:
- [Background] Yildirim P, Gultekin A, Yildirim A, Karahan AY, Tok F. Extracorporeal shock wave therapy versus corticosteroid injection in the treatment of trigger finger: a randomized controlled study. J Hand Surg Eur Vol. 2016 Nov;41(9):977-983. doi: 10.1177/1753193415622733. Epub 2016 Sep 28. PMID 26763271
- [Background] Nadar MS. Orthosis vs. exercise for the treatment of adult idiopathic trigger fingers: A randomized clinical trial. Prosthet Orthot Int. 2024 Dec 1;48(6):713-719. doi: 10.1097/PXR.0000000000000294. Epub 2023 Oct 20. PMID 37870373
- [Background] Teo SH, Ng DCL, Wong YKY. Effectiveness of proximal interphalangeal joint-blocking orthosis vs metacarpophalangeal joint-blocking orthosis in trigger digit management: A randomized clinical trial. J Hand Ther. 2019 Oct-Dec;32(4):444-451. doi: 10.1016/j.jht.2018.02.007. Epub 2018 Jul 18. PMID 30030005
- [Background] Chen YP, Lin CY, Kuo YJ, Lee OK. Extracorporeal Shockwave Therapy in the Treatment of Trigger Finger: A Randomized Controlled Study. Arch Phys Med Rehabil. 2021 Nov;102(11):2083-2090.e1. doi: 10.1016/j.apmr.2021.04.015. Epub 2021 May 21. PMID 34029555
- [Background] Vahdatpour B, Momeni F, Tahmasebi A, Taheri P. The Effect of Extracorporeal Shock Wave Therapy in the Treatment of Patients with Trigger Finger. Open Access J Sports Med. 2020 Mar 9;11:85-91. doi: 10.2147/OAJSM.S232727. eCollection 2020. PMID 32210646
- [Background] Gil JA, Hresko AM, Weiss AC. Current Concepts in the Management of Trigger Finger in Adults. J Am Acad Orthop Surg. 2020 Aug 1;28(15):e642-e650. doi: 10.5435/JAAOS-D-19-00614. PMID 32732655
- [Background] Tarbhai K, Hannah S, von Schroeder HP. Trigger finger treatment: a comparison of 2 splint designs. J Hand Surg Am. 2012 Feb;37(2):243-9, 249.e1. doi: 10.1016/j.jhsa.2011.10.038. Epub 2011 Dec 20. PMID 22189188